CLINICAL TRIAL: NCT02048865
Title: Apixaban for the Prevention of Venous Thromboembolism in High-Risk Ambulatory Cancer Patients: A Randomized Placebo-Controlled, Double-Blind Clinical Trial
Brief Title: Apixaban for the Prevention of Venous Thromboembolism in Cancer Patients
Acronym: AVERT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OHSN-20130563-01H; CV185-245 (Other Grant/Funding Number: Bristol-Myers Squibb)
Record Dates: First submitted 2014-01-27; First posted 2014-01-29 (Estimated); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Venous Thromboembolism; Cancer
Keywords: VTE Cancer
MeSH Terms: conditions — Venous Thromboembolism; Neoplasms | interventions — apixaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apixaban (Active Comparator): 2.5 mg BID for 6 months
  Interventions: Drug: Apixaban
- Placebo drug (Placebo Comparator): 2.5 mg BID for 6 months
  Interventions: Drug: Placebo drug

INTERVENTIONS:
Drug: Apixaban — Apixaban 2.5 mg tablets BID for 6 months
  Other Names: Eliquis
  Arms: Apixaban
Drug: Placebo drug — placebo drug 2.5mg BID for 6 months
  Arms: Placebo drug

SUMMARY:
Cancer patients have an increased risk of developing blood clots in the veins compared to non-cancer patients. Cancer patients who develop blood clots can lead to reduced life expectancy, delayed cancer treatment, and decreased quality of life. Prevention is the most effective way to decrease the complications associated with blood clots in the veins. Although previous clinical trials have shown some benefit on the use of medication to prevent blood clots in the veins in ambulatory cancer patients, these studies have been inconclusive in demonstrating that existing blood thinners significantly reduce the rate of blood clots in cancer patients. One possible explanation relates to the fact that these studies have included a large proportion of cancer patients who are a low risk of developing blood clots in the veins. We are proposing to identify cancer patients who are at a high risk of developing blood clots by using a validated tool at the time of their cancer diagnosis. The identified high risk cancer patients will be asked to participate in a trial to test the safety and efficacy of a new oral medication that has been used to prevent blood clots in patients undergoing surgery. We are enrolling 574 patients in 7 Canadian centers (Ottawa, Halifax, Montreal, Vancouver, Sault Ste. Marie, Toronto and Hamilton). 287 patients will receive the study drug and 287 will receive an inactive substance. Analysis will be performed to assess the safety and the superiority of the study drug.

DETAILED DESCRIPTION:
Patients holding a malignancy have a 7 to 28-fold higher risk for venous thromboembolism (VTE) than non-cancer patients(1). Since most cancer patients are currently treated in the outpatient setting, an acute episode of VTE has important implications on their care due to its effects on reduced life expectancy, high rates of VTE recurrence, therapeutic failures, delays in chemotherapy and the risk of bleeding during anticoagulation.

The best treatment of an acute episode of VTE is its prevention (thromboprophylaxis). Although previous clinical trials have shown some benefit on the use of thromboprophylaxis in ambulatory cancer patients, these studies have been inconclusive to convincingly demonstrate that existing anticoagulants significantly reduce the rate of VTE in cancer patients. Possible explanations are related to the fact that these studies have included a large number of cancer patients whose risk for VTE has been low and in consequence, the benefit of anticoagulation has become diluted by the large proportion of low risk cancer patients.

To increase the success of thromboprophylaxis in cancer outpatients, we propose, first, to include validated methods for predicting the risk of VTE at the time of cancer diagnosis(2, 3). This strategy will facilitate to identify cancer patients at high-risk for VTE and then, optimize the risk-to benefit ratio with anticoagulation. Second, to assess safety and efficacy of new oral anticoagulants in cancer patients as they represent an attractive alternative for an extended use of thromboprophylaxis. As a choice, new oral agents can be administered in fixed doses, do not require laboratory monitoring, have minimal interaction with additional drugs and provide a pain free alternative in patients who require injections.

Reference List

1. Blood Coagul Fibrinolysis 2011. Blood Coagul Fibrinolysis 2011;22:86-91.
2. Blood 2010. Blood 2010;116:5377-5382.
3. Blood 2008. Blood 2008;111:4902-4907.

ELIGIBILITY:
Inclusion Criteria:

* A newly diagnosed cancer site or progression of the malignant disease after complete or partial remission.
* Initiating a new course of chemotherapy with a minimum intent of 3 months therapy
* A VTE risk stratification score of ≥ 2, according to the scoring method
* Age 18 years old or older
* Provide written informed consent

Exclusion Criteria:

* Lesions or conditions at increased risk of clinically significant bleeding (eg. active peptic ulcer disease)
* Objectively confirmed substantial liver insufficiency as defined by clinical manifestations of ascites, cirrhosis, encephalopathy and/or jaundice and/or biochemical abnormalities in liver function tests including hypoalbuminemia (< 3.5 gr/dL), elevated levels of total bilirubin (> 25 umol/L), elevated liver transaminases (2 times the upper limit of normal) and/or biochemical diagnosis of biliary tract obstruction (elevated levels of gamma-glutamyl transferase and alkaline phosphatase, 3 times the upper limit of normal). *
* Diagnosis of basal cell or squamous cell carcinoma of the skin or acute leukemia or myelodysplastic syndrome**
* Planned stem cell transplant
* Life expectancy less than 6 months
* Acute or chronic renal insufficiency with glomerular filtration rate (GFR) < 30 ml/min calculated by the Cockroft and Gault formula.
* Pregnancy***
* Continuous anticoagulation with vitamin K antagonists, low-molecular-weight heparin (LMWH), or other oral anticoagulants
* Weight < 40 Kg
* Platelet count < 50 x 109/L
* Known allergies to ingredients contained in apixaban
* Use of any contraindicated medications with apixaban

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 575 (Actual)
Dates: Start 2014-03-24 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-19 (Actual)

PRIMARY OUTCOMES:
first episode of objectively documented, symptomatic or asymptomatic VTE (DVT and/or PE) | 7 months

SECONDARY OUTCOMES:
Rate of adverse events | 7 months
  rate of clinical overt bleeding( major and minor bleeding) and death within the study period

CONTACTS AND LOCATIONS:
Overall Officials: Phil Wells, MD, Principal Investigator — Ottawa Hospital Research Institute; Marc Carrier, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (14):
- Canada (14):
  - Vancouver General Hospital, Vancouver, British Columbia
  - Capital District Health Authority, Halifax, Nova Scotia
  - Royal Victoria Regional Health Centre (RVH), Barrie, Ontario
  - William Osler Health System -Brampton, Brampton, Ontario
  - Juravinski Hospital & Cancer Centre, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Center, London, Ontario
  - Lakeridge Health -Oshawa, Oshawa, Ontario
  - Ottawa Hospital-General Campus, Ottawa, Ontario
  - Sault Area Hospital, Sault Ste. Marie, Ontario
  - Markham Stouffville Hospital, Toronto, Ontario
  - Centre intégré de santé et de services sociaux de l'Outaouais - Gatineau, Gatineau, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Centre intégré de santé et de services sociaux du Bas St Laurent -Rimouski, Rimouski, Quebec

REFERENCES:
- [Derived] Brandt W, Brown C, Wang TF, Tagalakis V, Shivakumar S, Ciuffini LA, Mallick R, Wells PS, Carrier M. Efficacy and safety of apixaban for primary prevention of thromboembolism in patients with cancer and a central venous catheter: A subgroup analysis of the AVERT Trial. Thromb Res. 2022 Aug;216:8-10. doi: 10.1016/j.thromres.2022.05.014. Epub 2022 May 29. PMID 35660801
- [Derived] Wang TF, Mallick R, Carrier M, Wells PS. Safety and efficacy of apixaban thromboprophylaxis in ambulatory cancer patients according to renal function: A subgroup analysis of the AVERT trial. Thromb Res. 2022 Mar;211:85-87. doi: 10.1016/j.thromres.2022.01.022. Epub 2022 Jan 31. PMID 35124234
- [Derived] Kahale LA, Matar CF, Tsolakian I, Hakoum MB, Barba M, Yosuico VE, Terrenato I, Sperati F, Schunemann H, Akl EA. Oral anticoagulation in people with cancer who have no therapeutic or prophylactic indication for anticoagulation. Cochrane Database Syst Rev. 2021 Oct 8;10(10):CD006466. doi: 10.1002/14651858.CD006466.pub7. PMID 34622445
- [Derived] Ladha D, Mallick R, Wang TF, Caiano L, Wells PS, Carrier M. Efficacy and safety of apixaban for primary prevention in gastrointestinal cancers: A post-hoc analysis of the AVERT trial. Thromb Res. 2021 Jun;202:151-154. doi: 10.1016/j.thromres.2021.03.013. Epub 2021 Mar 21. PMID 33857789
- [Derived] Rutjes AW, Porreca E, Candeloro M, Valeriani E, Di Nisio M. Primary prophylaxis for venous thromboembolism in ambulatory cancer patients receiving chemotherapy. Cochrane Database Syst Rev. 2020 Dec 18;12(12):CD008500. doi: 10.1002/14651858.CD008500.pub5. PMID 33337539
- [Derived] Carrier M, Abou-Nassar K, Mallick R, Tagalakis V, Shivakumar S, Schattner A, Kuruvilla P, Hill D, Spadafora S, Marquis K, Trinkaus M, Tomiak A, Lee AYY, Gross PL, Lazo-Langner A, El-Maraghi R, Goss G, Le Gal G, Stewart D, Ramsay T, Rodger M, Witham D, Wells PS; AVERT Investigators. Apixaban to Prevent Venous Thromboembolism in Patients with Cancer. N Engl J Med. 2019 Feb 21;380(8):711-719. doi: 10.1056/NEJMoa1814468. Epub 2018 Dec 4. PMID 30511879